CLINICAL TRIAL: NCT05873062
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study of the Effects of Single Doses of AUT00201 in Patients With Myoclonus Epilepsy and Ataxia Due to Potassium (K+) Channel Mutation (MEAK)
Brief Title: Safety, Blood Levels and Effects of AUT00201 in Patients With MEAK
Acronym: AUT022201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: AUT022201
Record Dates: First submitted 2023-04-18; First posted 2023-05-24 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Myoclonus Epilepsies, Progressive
Keywords: MEAK; EPM7
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to one of the two treatments with 3-5 subjects per treatment sequence. Each subject will receive both treatments (100 mg AUT00201 and placebo) with a washout period of 1 day between single doses.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: AUT00201 (Experimental): Single dose (oral, capsule) of AUT00201
  Interventions: Drug: AUT00201
- Experimental: Placebo (Placebo Comparator): Single dose matching placebo oral capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUT00201 — Single oral dose
  Arms: Experimental: AUT00201
Drug: Placebo — Single oral dose
  Arms: Experimental: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, crossover study to assess the safety, tolerability, and pharmacokinetics of single doses of AUT00201 at 100 mg or matching placebo in patients with myoclonus epilepsy and ataxia due to potassium channel mutation (MEAK).

DETAILED DESCRIPTION:
6 to 10 patients aged 18 years and older, diagnosed with MEAK will be enrolled in the study. Patients will be administered a single dose of AUT00201 and matching placebo in a crossover design. The study is comprised of an outpatient screening and procedure orientation followed by approximately 5 days of an inpatient stay at a clinical research unit. After screening/orientation (Visit 1), and baseline assessments (Visit 2), patients will be administered a single dose of 100 mg of AUT00201 or matching placebo the morning of Visit 3. PK assessments will be done at Visits 3, 4, 5, and 6 from predose and up to 27 hours postdose. Visit 4 will be a washout day for patients. At Visit 5 patients will be administered the crossover treatment. At Visit 6 patients will be discharged from the unit. Safety and tolerability assessments will be conducted throughout. PD parameters will also be assessed. Patients will be followed up by telephone 14 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older at time of consenting.
* Diagnosed with MEAK, based on documented genetic evidence of the presence of the KCNC1 (c.959G>A; p.Arg320His) variant.
* If take anticonvulsants, must be on a stable anticonvulsant regiment for at least 30 days prior to Visit 1 and anticipated to remain stable throughout the study or if not on an anticonvulsant regimen, must be stable in regards to seizures for at least 30 days prior to Visit 1 and anticipated to remain stable throughout the study.
* Must be able to participate and willing to give written informed consent. If patient is unable to provide written informed consent, a legally authorized representative can sign on their behalf.
* Must be willing to perform study assessments and comply with the study protocol.
* If the patient is dependent on a caregiver and/or will need assistance either travelling to the site, whilst attending clinic visits and/or helping to document study assessment responses provided by the patient (eg, questionnaires administered on a tablet device), they must have an identified caregiver, considered reliable by the Investigator, to provide support to the patient for the duration of the study. The caregiver must be willing and able to provide support to the patient and, if required, stay for the duration of the study.
* Medically stable based on Investigator's judgement for at least 90 days prior to Visit 1.
* Women of childbearing potential must have a negative urine pregnancy test on Visit 2.
* If a vagal nerve stimulator is used, it must be implanted at least 150 days before Day. -1, and parameters must be stable for at least 30 days before Visit 1 and expected to remain stable throughout the study.
* If a ketogenic diet is followed, it must be stable for at least 30 days before Visit 1 and expected to remain stable throughout the study.
* Willing to comply with contraceptive requirements.
* Able to speak, read and understand English at a fluent level

Exclusion Criteria:

* Known pathogenic mutation in another gene that causes epilepsy or a different mutation in the KCNC1 gene than the c.959G>A variant.
* Clinically significant metabolic, hepatic, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder.
* Clinically significant abnormal vital signs or laboratory test results.
* Hypersensitivity to AUT00201 or any of the excipients.
* Any medical condition or other factors, as judged by the Investigator, which may interfere with the patient's participation in this study and/or compromise the patient's ability to safely complete the study.
* Known to abuse drugs or those who test positive on urine screen for drugs of abuse will be excluded based on Investigator's judgement.
* Positive hepatitis B surface antigen or hepatitis C antibody.
* Clinically significant abnormality on the 12-lead electrocardiogram.
* Having received an investigational product 90 days prior to Visit 1.
* Currently using felbamate <1 year prior to Visit 1, or any evidence of ongoing hepatic or bone marrow dysfunction associated with current/prior felbamate treatment. Patients who are currently using felbamate for >1 year prior to Visit 1 and have no evidence of ongoing hepatic or bone marrow dysfunction associated with felbamate treatment are allowed.
* Currently using vigabatrin and having received vigabatrin for <2 years prior to Visit 1.
* Suicidal ideation with some intent to act within 6 months prior to Visit 1 based upon response in the Columbia-Suicide Severity Rating Scale (positive response to questions 4 or 5 of the suicidal ideation section) and as judged by the Investigator as having a significant impact on trial participation or patient safety. History of suicidal behavior within 1 year prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gelfand, MD, Principal Investigator — Penn Epilepsy Center, Department of Neurology
Locations (1):
- University of Pennsylvania, Penn Epilepsy Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five unique patients were enrolled, however one patient was enrolled (signing two informed consent forms) and completed the study twice, in line with Protocol Amendment #3, resulting 6 participants being enrolled and completing the study. Six participants are reported for safety and PK data, the 5 unique are reported for baseline and demographics, and the numbers reported are indicated for each PD outcome.
Pre-assignment Details: All 6 participants who signed the informed consent form completed the study.
Groups:
- Experimental: AUT00201 / Placebo: Single dose of AUT00201 (oral, capsule) followed by a single dose of placebo to match
- Experimental: Placebo / AUT00201: Single dose of matching placebo (oral, capsule) followed by a single dose of AUT00201 (oral, capsule)
Period: Overall Study
Arm/Group | Experimental: AUT00201 / Placebo | Experimental: Placebo / AUT00201
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Placebo / AUT00201: Single dose matching placebo (oral, capsule) followed by a single dose of AUT00201 (oral, capsule)
- Total: Total of all reporting groups
Arm/Group | Experimental: AUT00201 / Placebo | Experimental: Placebo / AUT00201 | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events After Single Dose Treatment of AUT00201 Compared to Placebo
Time Frame: 19 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: AUT00201: Single dose of AUT00201 (oral, capsule)
- Experimental: Placebo: Single dose of matching placebo (oral, capsule)
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 6 | 6
Participants | 5 | 5

2. Secondary Outcome: Change From Baseline in Cortical Inhibition; as Measured by Paired-pulse Transcranial Magnetic Stimulation (ppTMS) at Short Interval Cortical Inhibition (SICI) Inter-stimulus-intervals (ISI): the Outcome is the Average %-Inhibition at SICI 2.5 and 3ms ISI
Description: ppTMS allows measurement of cortical inhibitory circuit functions. In ppTMS protocols 2 consecutive pulses are delivered to the hand motor region at a fixed interstimulus interval such that the motor-evoked potential, captured by surface EMG sensors, resultant from the second (test) stimulus is modulated by an conditioning stimulus. First resting motor threshold is recorded, which is defined as the lowest stimulus intensity (expressed as a percentage of maximal stimulator output, %MSO) required to induce motor evoked potentials of 50μV. SICI will be elicited with a conditioning stimulus of 70% of resting motor threshold at 2.5ms ISI and 3ms ISI. SICI at each ISI will be reported in %-inhibition and the average calculated for this outcome measure. An increase (positive change from baseline) would indicate a normalisation in this population. Post-dose collected 2-4h post dose on Day1 and Day3 (active vs placebo randomised crossover).
Time Frame: 2 - 4 hours post dose
Population: Modified Pharmacodynamic Population. Values reported are changes from baseline in the average SICI 2.5 and 3ms measurements from the 2 to 4 hour postdose assessment.
Measure: Mean (Standard Deviation); unit: % inhibition
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 3 | 3
% inhibition | 4.0300 (5.8674) | 4.0050 (8.6771)

3. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentrations (Cmax) of AUT00201
Time Frame: 27 hours
Population: No subjects analysed for PK parameters following the placebo dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Experimental: Placebo: Single dose matching placebo (oral, capsule)
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 6 | 0
ng/mL | 411 (273) |

4. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-time Curve (AUC) of AUT00201 to the Last Observed Quantifiable Concentration
Description: AUCt
Time Frame: 27 hours
Population: No PK parameters were analysed following placebo dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 6 | 0
ng*h/mL | 2110 (1170) |

5. Secondary Outcome: Change From Baseline in Measures of Dysarthria as Assessed by Speaking Rate Metric From Automated Standardized Speech Test.
Description: Baseline data were collected on Study Day -1 (V2); post-dose data were collected 1 hour post dose on Day 1 (V3) and Day 3 (V5) (active vs placebo randomised crossover).
  An increase (positive change from baseline) in syllables/sec would indicate an improvement in this population.
Time Frame: 1 hour post dose
Population: Modified Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: syllables/sec
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 4 | 5
syllables/sec | 0.7014 (0.6318) | 0.2161 (0.4487)

6. Secondary Outcome: Change From Baseline in Myoclonus Index (MI; a Measure of Positive Myoclonus) Evaluated With EMG and Accelerometer
Description: Average MI from 0 to 4 hours postdose, calculated during hourly finger-to-nose tasks and Unified Myoclonus Rating Scale Section 4 and 5 tasks, averaged across arms. The Myoclonus Index (MI) is a novel methodology for objectively measuring severity of positive myoclonus. The MI is calculated from positive myoclonus detected using surface electromyography (EMG) and accelerometry data, as described in the publication by Rissanen et al (Clin Neurophysiol. 2021).
  People who do not experience myoclonus would be expected to have a score of '0' on the Myoclonus Index; there is no maximum score, although higher scores indicate more severe myoclonus. A reduction of MI (negative change from baseline) would indicate an improvement in this population.
  Baseline data are collected on Study Day -1 (V2); post-dose data are collected hourly from dosing to 4 hours post dose, then averaged, on Day 1 (V3) and Day 3 (V5) (active vs placebo randomised crossover).
Time Frame: 0-4 hours post dose
Population: Modified Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 5 | 5
Index | 0.4556 (1.1175) | 0.4257 (1.0254)

7. Secondary Outcome: Change From Baseline in Measures of Dysarthria as Assessed by Buttercup Count From Automated Standardized Speech Test.
Description: Number of times the word "Buttercup" was correctly repeated within 30 seconds. An increase (positive change from baseline) in number of 'buttercups' would indicate an improvement in this population.
  Baseline data collected were collected on Study Day -1 (V2); post-dose data were collected 1-hour post-dose on Day 1 (V3) and Day 3 (V5) (active vs placebo randomised crossover).
Time Frame: 1 hour post-dose
Population: Modified Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Number correct "Buttercup"s in 30seconds
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
Number analyzed (Participants) | 3 | 4
Number correct "Buttercup"s in 30seconds | 0.0 (1.0) | -0.3 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events, based on clinical signs and symptoms and laboratory measurements, were collected from the time the ICF was signed until follow up phone call (end of study) Visit 7 (Study Day 18±2 days).
Arm/Group | Experimental: AUT00201 | Experimental: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: AUT00201 (N=6) | Experimental: Placebo (N=6)
Upper Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application Site Haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter Site Pain (General disorders) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Myoclonic Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT05873062/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT05873062/SAP_001.pdf